CLINICAL TRIAL: NCT03070860
Title: Glucidic Metabolism, Ossification and Arterial Calcification During PseudoXanthoma Elasticum (PXE)
Brief Title: What's Happen Under the Calcification Process in Pseudoxanthoma Elasticum
Acronym: GOCAPXE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-A01614-43
Record Dates: First submitted 2016-06-13; First posted 2017-03-06 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: Low Grade Chronic vascular and skin Inflammation; Molecular vascular and skin Calcification; Calcium Score
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Dermatitis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PXE Patient (Experimental): positron emission tomography scanner (PET scan) 18-FDG and 18-NAF: conventionnal use.
  Interventions: Radiation: PET scan 18-FDG and 18-NAF

INTERVENTIONS:
Radiation: PET scan 18-FDG and 18-NAF — Positron emission tomography (PET) is a medical imaging test performed in a nuclear medicine department.
  PET scan is performed by IV injection of a mildly radioactive tracer (NAF and FDG).
  Other Names: positron emission tomography

SUMMARY:
The investigators hypothesize is that in PXE patients, low grade chronic inflammation could preceed the molecular and the clinical calcification process.

DETAILED DESCRIPTION:
Pseudoxanthoma elasticum (PXE; OMIM 264800), is an autosomal recessive metabolic disorder characterized by the fragmentation and progressive calcification of elastic fibers(elastorrhexis) in connective tissue in the skin, Bruch's membrane of the retina and the vascular system. PXE is caused by mutations in the ABCC6 (ATP-binding cassette subfamily C member 6) gene, located on the short arm of chromosome 16, encoding a transmembrane ATP binding anion transporter normally expressed in the liver and the kidney. The pathophysiology of PXE, particularly the mechanism of ectopic mineralization, remains largely unknown. PXE is currently an intractable disease, associated with considerable morbidity and occasional mortality due to cardiovascular complications. The major symptoms of the disease are characterized by unaesthetic skin folds, central blindness and cardiovascular complication with an early and severe peripheral arterial disease (PAD) and complication at younger age than the normal population. Unfortunately, histological studies are limited by the availability of arterial tissue from patients but it has been showed calcium deposition in the media layer of the large (i.e. aorta, carotids and femoral) and medium sized vessels (i.e. radial and ankle arteries) (ref). However, the underlying pathophysiology for arterial calcification in PXE remains incompletely defined, and there are currently no effective medical treatments capable of altering its course.

No longitudinal study has been performed to explain the calcification process in PXE. As PXE is a systemic metabolic disease, low grade inflammation could be the trigger of a deregulated inflammation resolution process resulted in calcification. Thus, alternative techniques are therefore required to investigate the pathogenesis and progression of this condition.

Positron emission tomography (PET) combined with computed tomography (CT) is a noninvasive imaging technique that allows the identification and quantification of specific biochemical processes within small anatomic structures, such as vascular wall. Furthermore, 2 common PET tracers target calcification and inflammation, which are believed to play a key role in the development of the disease. 18F Flurodeoxyglucose (18F-FDG) is a glucose analogue that is taken up into cells by glucose transport proteins and enters the glycolytic metabolic pathway. After the initial hexokinase step, 18F-FDG-6-phosphate cannot be metabolized further and becomes trapped within cells that have high metabolic requirements, such as macrophages. PET imaging with the use of 18F-FDG has become an established means of quantifying vascular inflammation in both the aorta and carotid arteries, correlating with plaque macrophage burden and symptomatic status. 18F-Sodium fluoride (18FNaF) is an alternative PET tracer that is directly incorporated into exposed bone crystal (hydroxyapatite) via an exchange mechanism with hydroxyl groups. It is therefore thought to detect areas of novel calcification and regions of calcium remodeling and is used clinically for the detection of primary osteoblastic tumors and bone metastases. More recently, studies have described 18F-NaF uptake as a marker of calcification within atherosclerotic plaque. More recently, the calcifying process was examined in 4 PXE patients using 18NaF PET/CT showing in the femoral arteries, increased arterial wall 18NaF signal at levels similar to those for cortical bone. However, the mechanism responsible for the increased osteoblastic activity leading to arterial wall calcification in PXE remains unknown.

.

In this study, the investigators investigated 18F-NaF and 18F-FDG uptake in the arterial wall and skin of patients with PXE with 3 major aims: :

1. Does low grade inflammation in vascular wall and skin exist in PXE patient and a specificity site might exist?
2. Does low grade inflammation in vascular wall and skin quantified by 18F-FDG preceed the molecular calcification process quantified by 18F-NaF?
3. Does low grade inflammation and bone turn over correlate conversely to calcium score?

ELIGIBILITY:
Inclusion Criteria:

* PXE patient diagnosed according the international criteria
* Informed consent obtained
* Patient affiliated to Health care system

Exclusion criteria included inability or unwillingness to provide informed consent. Also, women of childbearing age not receiving contraception, pregnant women, nursing women, diabetic patients, patients with osteopenia, inflammatory or autoimmune systemic disease, high blood glucose concentrations (> 11 mmol/L) because of the competition between glucose and 18F-FDG for cellular entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Vascular Inflammation | 90min post injection : 1 time
  Measurement 18F-FDG TBRs of patients with PXE; and the comparison of 18F-NaF femoral arteries' TBRs with popliteal artery's TBRs of patients with PXE (at 30 min and 90min post injection).
Molecular Calcification | 90min post injection : 1 time
  Measurement 18F-NaF femoral arteries' TBRs with popliteal artery's TBRs of patients with PXE

CONTACTS AND LOCATIONS:
Overall Officials: Loukman OMARJEE, MD,MSc, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided